CLINICAL TRIAL: NCT05877235
Title: Serum Concentration of Endogenous Estrogens and Sirtuin-1 in Postmenopausal Women With Atherosclerotic Coronary Heart Disease After Administration of Atorvastatin and Supplementation With Quercetin: a Randomized Study
Brief Title: Serum Concentration of Endogenous Estrogens and Sirtuin-1 After Administration of Atorvastatin and Quercetin:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, ANTONIO DE PADUA MANSUR, Associate Professor, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64417922.0.0000.0068
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease; Menopause
Keywords: Coronary disease; Atherosclerosis; Estradiol; Estrone; Sirt1; Quercetin; Atorvastatin; Polyphenols
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Atherosclerosis | interventions — Quercetin

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial, parallel and placebo-controlled.
Who Masked: Participant, Care Provider
Masking Description: Participants in the control group will receive capsules identical to those in the intervention group, but with cornstarch.
  The care provider and the participants do not have the information about which capsules the participant is taking, and do not have access to which groups the patients belong. Statistical analyses will be performed on a blinded database, i.e. without information of which groups the participants belong to.
  Only the principal investigator of the study has this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quercetin (Experimental): Trans-quercetin, 1000 mg daily for 60 days
  Interventions: Dietary Supplement: Quercetin
- Atorvastatin (Experimental): Atorvastatin, 80mg daily for 60 days.
  Interventions: Dietary Supplement: Quercetin
- Control (Placebo Comparator): Starch, 1000mg daily for 60 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin — Trans-quercetin, 1000 mg daily for 60 days
  Arms: Atorvastatin; Quercetin
Dietary Supplement: Placebo — Starch, 1000 mg daily for 60 days
  Arms: Control

SUMMARY:
Chronic coronary syndrome (CCS) is the leading cause of death in women in the most developed regions of Brazil. The primary etiopathogenic mechanism is the process of atherosclerosis. A healthy diet rich in fruits and vegetables is associated with a lower incidence of CCS. The higher consumption of these foods promotes greater availability of phenolic compounds, and the higher intake of these compounds is one of the main hypotheses for vascular health. Quercetin, a phenolic compound, is the most abundant natural antioxidant belonging to the group of flavonoids. Quercetin improves lipoprotein metabolism, has an antioxidant capacity, produces vasodilating substances in the vascular endothelium, and reduces platelet aggregability. Likewise, statins are medications known to reduce cardiovascular events in women with CCS by reducing serum LDL-cholesterol levels and, to a lesser extent, by possible pleiotropic effects. In turn, SIRT1 is one of the 7 classes of proteins. It mediates various metabolic pathways in response to nutritional stimuli, particularly for caloric restriction and phenolic compounds, as well as coordinating the production and secretion of important hormones. However, the impact of quercetin supplementation and statin administration on serum endogenous estrogen levels is unknown

DETAILED DESCRIPTION:
The main objective of this study is to investigate the influence of atorvastatin and of quercetin in the serum concentrations of estradiol and estrone after the administration of atorvastatin and supplementation with quercetin. This is a randomized, double-blind, placebo-controlled, 60-day study in 60 postmenopausal women with CAD, divided into three groups of 20 women each: Group 1 - quercetin (500 mg/day); Group 2 - atorvastatin (80 mg/day); Group 3 - control (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women;
* Diagnosed coronary artery disease;
* Stable coronary disease;

Exclusion Criteria:

* hypo or hyperthyroidism,
* rheumatic disease,
* use of alcohol,
* hepatic failure,
* renal failure
* hormone replacement therapy
* use of insulin

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
Estradiol | 60 days
  serum concentrations
Estrone | 60 days
  serum concentrations
Sirtuin-1 | 60 days
  Serum concentrations and gene expression

SECONDARY OUTCOMES:
Cardiometabolic risk factors | 60 days
  Lipid and glucometabolic profiles

CONTACTS AND LOCATIONS:
Locations (1):
- INCOR- Heart Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No